CLINICAL TRIAL: NCT07371091
Title: Monitoring the Use of Collagen Dura Membrane - Repair (DMR) in the Post-market Phase
Brief Title: Post-market Clinical Investigation Plan: Collagen Dura Regeneration Membrane - Repair (DMR)
Status: Not yet recruiting | Type: Observational
Sponsor: Collagen Matrix (Industry)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP.088
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Repair of Dura Mater

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Monitoring the Use of Collagen Dura Regeneration Membrane - Repair (DMR) in the Post-market Phase.

DETAILED DESCRIPTION:
A multi-center (up to 4 sites) clinical case series of 110 patients treated with Collagen Dura Regeneration Membrane - Repair (DMR) for a dural defect in the dura mater will be evaluated prospectively. The primary endpoint is the rate of adverse events related to the Subject Device requiring surgical intervention. Patients will have a follow-up evaluation post-operatively in line with standard or care of the study site, and 8 months after the initial surgery. No original patient records or personal identifying information will be disclosed to CMI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a dural defect requiring repair with a dural substitute as per routine clinical practice
* Patient is 18 years or older
* Patient of child-bearing potential is not pregnant or nursing
* Participant is willing and able to provide consent

Exclusion Criteria:

* Patients with a known history of hypersensitivity to bovine derived materials
* Patients that are non-English speaking
* Patients requiring legal representation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a dural defect requiring repair with a dural substitute.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Revision Surgery | at least one timepoint at 8 months or more post-surgery
  Rate of adverse events related to the Subject Device requiring surgical intervention.

SECONDARY OUTCOMES:
Rate of Adverse Events | at least one timepoint at 8 months or more post-surgery
  Intra-operative and post-operative adverse events (i.e., infection, CSF Leak, and Pseudomeningocele)
Product Performance | at least one timepoint at 8 months or more post-surgery
  Score of adequacy of product performance - 1 (poor) to 4 (excellent)
Product Handling at Implantation | Initial surgery
  Score for product handling at implantation - 1 (poor) to 4 (excellent)
Product Adaptability at Implantation | Initial surgery
  Score for product adaptability at implantation - 1 (poor) to 4 (excellent)